CLINICAL TRIAL: NCT03979794
Title: A Distress Screening and Intervention in Cancer Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient funding for research personnel prevented adequate recruitment and retention of research participants.
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Chelsea Ratcliff, Adjunct Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-40276
Record Dates: First submitted 2019-05-28; First posted 2019-06-07 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Cancer; Stress
MeSH Terms: conditions — Neoplasms | interventions — Behavior Therapy; Health

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial (intervention vs. standard care)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Be-WEL Intervention (Experimental): Behavioral Intervention for Wellness and Engaged Living (Be-WEL) is a 4-session (2 preoperative, 2 postoperative) telephone intervention focused on improving emotional and physical health through relaxation, behavioral activation, increased physical activity, and adherence to medication and wound care.
  Interventions: Behavioral: Behavioral Intervention for Wellness and Engaged Living (Be-WEL)
- Standard Care (No Intervention): Standard Care consists of the standard care patients typically receive from their medical team.

INTERVENTIONS:
Behavioral: Behavioral Intervention for Wellness and Engaged Living (Be-WEL) — Behavioral Intervention for Wellness and Engaged Living (Be-WEL) is a 4-session (2 preoperative, 2 postoperative) telephone intervention focused on improving emotional and physical health through relaxation, behavioral activation, increased physical activity, and adherence to medication and wound care.
  Arms: Be-WEL Intervention

SUMMARY:
The goal of this project is to examine initial effectiveness of a brief (2 preoperative, 2 postoperative session) cognitive behaviorally-based telephone intervention compared to standard care on postoperative outcomes for patients who are scheduled to undergo a cancer-related surgery in 12 or more days and screen positive for distress (4 or higher on 0-10 Distress Thermometer). The intervention focuses on improving emotional and physical health through relaxation, behavioral activation, increased physical activity, and adherence to medication and wound care. Participants will be randomly assigned to receive the intervention or to receive standard care. Outcomes assessed 4 and 6 weeks post-operatively will include: Depression (Patient Health Questionnaire-8), anxiety (Generalized Anxiety Disorder-7), health-related QOL (SF-36 MCS and PCS), number and type of complications, length of stay, and 30-day readmission.

ELIGIBILITY:
Inclusion Criteria:

* ADULT (18 years of age or older)
* SCHEDULED FOR SURGERY FOR CANCER (excluding non-melanoma skin cancer) 12 OR MORE DAYS IN ADVANCE OF CONSENT
* SIGNIFICANTLY DISTRESSED (>4 on the 0-10 Distress Thermometer)
* ABLE TO SPEAK ENGLISH

Exclusion Criteria:

* COGNITIVE IMPAIRMENT : <4 on baseline Mini Cog measure
* SERIOUS MENTAL ILLNESS: a diagnosis of a bipolar or psychotic disorder (noted in medical record)
* NON-ENGLISH SPEAKING: This study only involves participants who can speak English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2024-11-12 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-8 | 4-weeks post-operation (+/-1 week)
  PHQ-8 assesses depression symptoms; A total score (range: 0-24) will be used with higher scores representing more depressive symptoms.
Generalized Anxiety Disorder-7 | 4-weeks post-operation (+/-1 week)
  The GAD-7 measures anxiety symptoms; A total score (range: 0-21) will be used with higher scores representing more anxiety symptoms.

SECONDARY OUTCOMES:
Medical Outcomes Study Short Form-36 (SF-36) Physical Health Component Scale (PCS) | 4-weeks post-operation (+/-1 week)
  The SF-36 PCS assesses physical health-related quality of life (QOL) on a 0-100 scale (with a mean of 50 and standard deviation of 10 for general population). Higher scores represent higher physical health-related QOL.
Medical Outcomes Study Short Form-36 (SF-36) Mental Health Component Scale (MCS) | 4-weeks post-operation (+/-1 week)
  The SF-36 MCS assesses mental health-related quality of life (QOL) on a 0-100 scale (with a mean of 50 and standard deviation of 10 for general population). Higher scores represent higher mental health-related QOL.
Number of Complications | 30 days post-operation
  Occurrence of: perioperative mortality, cardiac complications, postoperative pneumonia, intubation for >48-hours postoperatively unplanned reintubation, venous thromboembolic events, renal dysfunction, or surgical-site infections
Length of post-operative hospital stay | 30 days post-operation
  Number of days inpatient hospital stay after operation
Hospital Readmission | 30 days post-operation
  Number of times readmitted to a hospital after operation

CONTACTS AND LOCATIONS:
Overall Officials: Chelsea G Ratcliff, PhD, Principal Investigator — Baylor College of Medicine/Sam Houston State University
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
There is not currently a plan to make individual participant data available to other researchers.